CLINICAL TRIAL: NCT02093754
Title: Assessing the Severity of Metabolic-related Liver Injuries in Aging HIV-monoinfected Patients: a European Multicentre Study
Brief Title: Assessing the Severity of Metabolic-related Liver Injuries in Aging HIV-monoinfected Patients
Acronym: ANRS ECHAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ECHAM; 2012-A01670-43 (Other: Competent authority ANSM)
Record Dates: First submitted 2014-01-17; First posted 2014-03-21 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: HIV Infection; Liver Injuries
MeSH Terms: conditions — HIV Infections | interventions — Magnetic Resonance Spectroscopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: MRI and biopsy

SUMMARY:
This study will allow to assess liver related injuries in HIV patients.

DETAILED DESCRIPTION:
This study is a cross-sectional, multicentre study including 7 centres from 3 European countries (Belgium, France, Germany).

The maximum duration of the study for each patient will be 4 months, consisting of:

* a screening visit,
* an inclusion visit to perform the biologic tests and exams necessary for the study, within 1 month after the screening visit,
* a result delivery visit within 1 month after inclusion visit, to disclose results of previous investigations. Patients with one or two non invasive markers suggesting significant fibrosis (≥F2) will be invited for liver biopsy within the next 2 months.
* a "liver biopsy" visit, within 2 months after visit 2, liver biopsy in selected and consented patients

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥40 years
2. Infection with HIV-1
3. Cumulative exposure to cART for at least 5 years and currently under cART
4. Viral load < 400 copies/mL
5. CD4 count > 100 CD4/mm3
6. Female may be eligible to enter and participate in the study if she:

   * is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or
   * is of child-bearing potential with a negative blood pregnancy test at screening visit
7. Informed consent signed prior to any study procedure
8. To be covered by a medical insurance (only for French centres)
9. Presence of:

   * the metabolic syndrome as defined by the most recent international consensus definition (Alberti et al. Circulation 2009) including three components among the following criteria:

     * visceral obesity (waist circumference: Europeans and Africans ≥ 94 cm for men and ≥ 80 cm for women, Americans ≥ 102 cm for men and ≥ 88 cm for women, Asians ≥ 90 cm for men and ≥ 80 cm for women)
     * blood glucose ≥ 1 g/L (5,6 mmol/L) or anti-diabetic treatment,
     * serum triglycerides ≥ 1,5 g/L (1,7 mmol/L) or hypertriglycerides treatment,
     * serum HDL cholesterol < 0,4 g/L (1 mmol/L) for men and < 0,5 g/L (1,3 mmol/L) for women or hypercholesterolemia treatment,
     * blood pressure (Diastolic ≥130 mmHg and/or Systolic ≥ 85 mmHg) or antihypertensive treatment
   * and/or clinical lipoatrophy and/or lipohypertrophy using clinical questionnaires used and validated in previous published studies (ANRS 121 Hippocampe trial),
   * and/or chronic elevated transaminases ≥ 1.5 ULN and / or GGT ≥ 2 ULN confirmed by two blood samples within at least three-month interval over twelve months prior screening visit.

Exclusion Criteria:

1. Coinfection with hepatitis B (positive HBs antigen or isolated positive HBc antibody with positive PCR)
2. Positive HCV serology
3. Coinfection HIV-1 and HIV-2
4. Use of intravenous drugs within the last six months
5. Excessive alcohol intake (male > 50 g/d, female > 40 g/d)
6. Other causes of liver diseases i.e: viral hepatitis, hemochromatosis, Wilson disease, autoimmune hepatitis, primary or secondary biliary cirrhosis, primary or secondary cholangitis, α1 antitrypsine deficiency
7. Other causes of liver steatosis: current steroid therapy, current therapy with amiodarone, tamoxifen, methotrexate, nifedipine, or hycanthone; history of cancer chemotherapy; short bowel syndrome, polycystic ovarian syndrome, Weber-Christian disease
8. Active opportunistic infection except for candida oesophagitis
9. Current Cancer
10. Pregnancy
11. Decompensated heart failure
12. Subject under legal guardianship
13. Inability to give informed consent or incapacitation
14. Contra-indication to MRI: pace-maker, neurovascular surgery, intraocular materials, cochlear implant, severe claustrophobia
15. Participation in another study with an ongoing exclusion period at screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Percentage of steatosis detected by MRI | Within 6 months after all patients have completed MRI

SECONDARY OUTCOMES:
Percentage of fibrosis or cirrhosis using non invasive markers and concordance of non invasive markers | Within 6 months after all patients have completed the study
Risk factors (age, duration of infection, treatment, clinical and biological metabolic and adipose tissue parameters) of liver injuries | Within 6 months after all patients have completed the study
Independent risk factors of NAFLD, NASH and fibrosis (including markers of insulin resistance, inflammatory cytokines, markers of immune activation, adipokines) | Within 6 months after all patients have completed the study
Establish a diagnosis score based on biomarkers of liver injuries (Adiponectin, leptin, IL6, CRP, CD14) | Within 6 months after all patients have completed the study
  Quantifiable levels of serum adiponectin, serum leptin, serum HS-IL-6, HS-CRP, serum s-CD14 will be measured.
Description of pathogenetic factors and correlates with autophagy in liver biopsies of patients with evidence for liver fibrosis | Within 6 months after all patients have completed the study
  Autophagosome formation in the liver biopsies (only for patients presenting liver fibrosis equal or > 2 will be quantified.
Identification of features of the adaptive immune system associated to NAFLD, NASH and fibrosis (T cell activation, surface expression of Treg, NK cells, NKT cells) | Within 6 months after all patients have completed the study
  Quantifiable levels of T cell activation (in PBMC), Frequency and phenotype of Tregs (in PBMC), Quantifiable levels of NK cells (in PBMC), Quantifiable levels of Th17 and γδ T cell (in PBMC), Quantifiable levels of Plasma LPS and LPB (sCD163, CD26, Cytokeratin 18) will be measured.
Impact of IL28B and PNPLA3 genetic polymorphisms on the severity of liver steatosis, inflammation and fibrosis | Within 6 months after all patients have completed the study
Percentage of patients with NASH, fibrosis and cirrhosis on liver biopsy | Within 6 months after all patients have completed the study

CONTACTS AND LOCATIONS:
Overall Officials: Maud LEMOINE, MD, Principal Investigator — Medical Research Council
Locations (7):
- CHU Brussels, Brussels, Belgium
- France (2):
  - Hôpital la Salpêtrière, Paris
  - Hôpital Saint Antoine, Paris
- Germany (4):
  - Medical Center for Infectious Diseases, Berlin
  - Center for HIV and Hepato-Gastroenterology, Düsseldorf
  - University Medical Center, Hamburg
  - Hannover Medical School, Hanover